CLINICAL TRIAL: NCT06141980
Title: A Multi-center, phase3, Open-label Study to Evaluate the Long Term Safety and Efficacy of DWP16001 in Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin and Gemigliptin
Brief Title: Study to Evaluate the Long Term Safety and Efficacy of DWP16001 in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001308
Record Dates: First submitted 2023-11-10; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Enavogliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (DWP16001 0.3 mg) (Experimental): DWP16001 0.3mg, Tablets, Orally, Once daily
  Interventions: Drug: DWP16001 0.3 mg

INTERVENTIONS:
Drug: DWP16001 0.3 mg — DWP16001 0.3mg, Tablets, Orally, Once daily

SUMMARY:
The subjects, having voluntarily agreed to participate in the clinical trial and provided informed consent, will undergo screening tests. During Visit 1 (Screening), subjects meeting the inclusion/exclusion criteria will go through an 8-week stabilization period.

At Visit 1-1, central laboratory tests will be conducted. If the test results meet the criteria for Visit 2 (Enrollment Visit), the subject will be eligible to participate in the clinical trial.

The subjects will receive the investigational drug (DWP16001 0.3 mg) once a day for 52 weeks. They will visit the clinical trial site at weeks 8, 16, 24, 38, and 52 for safety and efficacy assessments during the 52-week treatment period.

DETAILED DESCRIPTION:
The subjects, having voluntarily agreed to participate in the clinical trial and provided informed consent, will undergo screening tests. During Visit 1 (Screening), subjects meeting the inclusion/exclusion criteria will go through an 8-week stabilization period. Throughout this period, subjects will receive concurrent administration of metformin (≥1,000 mg/day) and gemigliptin (50 mg/day), and will have a washout period for other oral antidiabetic drugs.

At Visit 1-1, central laboratory tests will be conducted. If the test results meet the criteria for Visit 2 (Enrollment Visit), the subject will be eligible to participate in the clinical trial.

The subjects will receive the investigational drug (DWP16001 0.3 mg) once a day for 52 weeks. They will visit the clinical trial site at weeks 8, 16, 24, 38, and 52 for safety and efficacy assessments during the 52-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with T2DM age 19 ~ under 80 years
2. Subjects who have 7% ≤ HbA1c ≤ 11% in screening visit(V1-1)
3. Subjects who have FPG <270 mg/dl screening visit(V1-1)
4. Subjects who have received a combination of metformin (≥1,000 mg/day) and gemigliptin (50 mg/day) for a minimum of 8 weeks prior to Visit 2 (Enrollment Visit)
5. Subjects who voluntarily decided to participate and provided written consent after being told of the objectives, method, and effects of this study

Exclusion Criteria:

1. Subjects with current or history of hypersensitivity to the IP of this study, metformin or drugs of the same class and their components (e.g., history of hypersensitivity to biguanide or SGLT2 inhibitors)
2. Diabetic ketoacidosis, diabetic coma or precoma within the past year
3. Urinary tract infections or genital infections within
4. Uncontrolled hypertension (SBP > 180 mmHg or DBP > 110 mmHg)
5. eGFR < 45 mL/min/1.73 m2
6. Severe heart failure (NYHA class III/IV

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety outcomes_Adverse events occurred during clinical trials | from baseline up to 52 weeks
  Safety outcomes_Adverse events occurred during clinical trials
Safety outcomes_ Change of blood pressure | from baseline to Week 8, 16, 24, 38, and 52 after administration of the IP
  Safety outcomes_ Change of blood pressure
Safety outcomes_ Change of heartbeat | from baseline to Week 8, 16, 24, 38, and 52 after administration of the IP
  Safety outcomes_ Change of heartbeat
Safety outcomes_ Change of body temperature | from baseline to Week 8, 16, 24, 38, and 52 after administration of the IP
  Safety outcomes_ Change of body temperature
Efficacy outcome_Change of HbA1c | from Baseline at Week 8, 16, 24, 38, and 52 after administration of the IP
  Efficacy outcome_Change of HbA1c
Efficacy outcome_Change of FPG | from baseline at Week 8, 16, 24, 38, and 52 after administration of the IP
  Efficacy outcome_Change of FPG
Efficacy outcome_Proportion of subjects achieving HbA1c target of < 6.5% | at Weeks 8, 16, 24, 38 and 52 after administration of the IP
  Efficacy outcome_Proportion of subjects achieving HbA1c target of < 6.5%
Efficacy outcome_Proportion of subjects achieving HbA1c target of < 7.0 % | at Weeks 8, 16, 24, 38 and 52 after administration of the IP
  Efficacy outcome_Proportion of subjects achieving HbA1c target of < 6.5%

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PH.D, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No